CLINICAL TRIAL: NCT02695953
Title: Neurobiology of Posttraumatic Stress Disorder Dysfunction and Recovery Following Cognitive Processing Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Milissa Kaufman (Other)
Responsible Party: Sponsor-Investigator, Milissa Kaufman, Medical Director, Hill Center for Women, Mclean Hospital
Organization: Mclean Hospital (Other)
Other Study IDs: 2015P001812
Record Dates: First submitted 2016-02-11; First posted 2016-03-02 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; biomarker; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Posttraumatic stress disorder (PTSD) is a significant personal and societal burden. The purpose of this study is to examine genetic, epigenetic, behavioral, and brain activity changes related to PTSD dysfunction and recovery before and after treatment with Cognitive Processing Therapy.

DETAILED DESCRIPTION:
Using functional magnetic resonance imaging approaches, the present research aims to examine the relationship between traumatic experience and the neural mechanisms of various PTSD symptoms, and determine how this relationship changes during PTSD extinction. Also, this proposal aims to better understand how the genetic/epigenetic profile of several genes predicts, and perhaps changes, in response to recovery from PTSD along with its neural correlates. This understanding will help identify individuals who will respond most optimally to a specific empirically based PTSD treatment, Cognitive Processing Therapy, while further connecting genetic biomarkers of risk with neural intermediate phenotypes underlying PTSD symptomatology.This study is observational as the investigator does not assign specific interventions to the participants of the study.

ELIGIBILITY:
Inclusion Criteria:

* PTSD diagnosis, as measured by the Clinician Administered PTSD Scale for DSM-5
* history of chronic childhood trauma due to relational abuse
* Ability to understand and sign informed consent
* Enrollment in CPT program at McLean Hospital
* Both genders, all ethnic backgrounds, age between 18 and 55
* Fluent English speakers
* Normal or Corrected Vision

Exclusion Criteria:

* History or current schizophrenia spectrum disorder or other psychotic disorders
* History or current bipolar or other related disorders
* Alcohol and/or substance use disorder within the past month
* Metal implants
* Medical or neurological illness (e.g., seizures, head injury in which they experienced a loss of consciousness)
* Positive pregnancy test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will include 102 individuals (half female) between the ages of 18 and 55 with a current diagnosis of PTSD as measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5). Participants must have a history of chronic childhood trauma due to relational abuse. All participants will be recruited from the McLean Hospital outpatient trauma track Cognitive Processing Therapy (CPT) treatment program.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2016-03; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Potential Change in Evidence of PTSD symptoms with neuroimaging | Within 30 days before and again within 30 days after Cognitive Processing Therapy Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Milissa L Kaufman, MD/PhD, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided